CLINICAL TRIAL: NCT04760223
Title: Reducing Depression-related Stigma and Increasing Treatment-seeking Among Adolescents: Randomized Controlled Trial of a Brief Video Intervention
Brief Title: Reducing Stigma Towards Depression Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, NYSPI, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ResearchFMH
Record Dates: First submitted 2021-02-11; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Stigma, Social
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video intervention 1 (Experimental): We presented a 100-second video to study participants to reduce stigma towards depression (a boy presenter). The protagonist discussed his own depression and how getting help assist him.
  Interventions: Behavioral: Video intervention
- Video intervention 2 (Experimental): We presented a 100-second video to study participants to reduce stigma towards depression (a girl presenter). The protagonist discussed his own depression and how getting help assist her.
  Interventions: Behavioral: Video intervention
- control video 1 (Placebo Comparator): A 100-second video presenting a boy without depression
  Interventions: Behavioral: Video intervention
- control video 2 (Placebo Comparator): A 100-second video presenting a girl without depression
  Interventions: Behavioral: Video intervention

INTERVENTIONS:
Behavioral: Video intervention — a 100-second video, presenting a personal story of a boy/girl dealing with depression

SUMMARY:
The investigators conducted a randomized controlled study to test the utility of a brief video-based intervention to: 1) reduce stigma towards depression, and 2) increase treatment-seeking intentions among adolescents.

DETAILED DESCRIPTION:
Young people present with the higher prevalence of mental health disorders compared to individuals at any other age, with up to 20% of adolescents likely to experience mental health disorders. Around 50% of mental health conditions start before the age of 14 and the onset of 75% of cases is before the age of 18. Depression is the most common diagnosis and epidemiological studies suggest that at any one time 8% to 10% of adolescents have severe depression. This means that the major burden of assessing and managing adolescent depression falls on primary care practitioners. Depression is a principal cause of illness and disability in teenagers, and suicide is the third most common cause of death among older adolescents. Mental health problems can significantly affect the development of children and young people having an enduring impact on their health and social functioning in adulthood. However, 75% of adolescents with mental health problems are not in contact with mental health services,8 and the primary reason for the reluctance to seek help is stigma.

Stigma refers to negative beliefs and stereotypes held toward a specific group of people and adversely affects people with mental illness. Public stigma refers to negative attitudes and beliefs that motivate individuals to fear, reject, avoid, and discriminate against people with mental illness. Individuals with mental illness expect to face prejudice and discrimination (anticipated stigma) and internalize public stereotypes of people with mental illness (self-stigma). Adolescents are particularly aware of how others perceive them and care greatly about what their peers think of them. Public stigma toward youngsters with mental illness has been identified as a barrier to seeking help; therefore, reducing public stigma among young people at risk for or even experiencing depression could enhance their receptivity to seeking help or treatment.

Applying strategies to reduce stigma towards mental health care among adolescents with high levels of depression may prevent worsening of symptoms, ameliorate impaired functioning, and reduce risks for long-term psychiatric illness. Among possible strategies, studies19 have shown that social contact is the most effective type of intervention to reduce stigmatizing attitudes. Social contact involves interpersonal contact with members of the stigmatized group: members of the general public who meet and interact with individuals who suffer from depression are likely to lessen their stigma. Corrigan identified the most important ingredients of contact-based programs: an empowered presenter with lived experience who attains his/her goals (e.g., "I was able to fight the depression and go back to school"). Although direct, in-person social contact, as well as indirect, video-based social contact have effectively improved attitudes toward mental issues and care, the latter can be implemented on a larger scale, use minimal resources and be easily disseminated.

The purpose of this study is to: (1) examine adolescents' stigma-related attitudes towards depression; and (2) test the utility of a brief video-based intervention in reducing stigma towards depression and increasing help-seeking intentions.

The investigators propose to randomly assign 1,000 individuals aged 14-18 in to either: (a) brief video-based intervention 1 ('Video 1'); (b) brief video-based intervention 2 ('Video 2'); or (c) no intervention video control arm ('Control'). The intervention videos will focus on empowered presenters with depression. The presenters will be 16-year-old adolescent professional actors, one of them is a boy (Video 1), one is a girl (Video 2). They each will share his/her personal story regarding depression and describe how social support from family, friends, and professionals have helped them overcome their symptoms and recover. The third group will watch a same length video with unrelated contents. Assessments will occur at baseline and at post-intervention and will tap into demographic identifiers and attitudes around stigma and help-seeking questionnaires.

Actors will be hired through the Child Study Center, and / or through the Standardized Patient Program of Teaching and Learning Center, Yale School of Medicine. Actors will be compensated and follow standardized patient best practices, including those specifically pertaining to under-age actors.

ELIGIBILITY:
Inclusion Criteria:

* 14-18-year-old
* US residents
* English speaker

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1183 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Stigma levels | Through the study completion (pre and post-intervention), an average of one month
  Level of stigma towards depression measured by the 9-item Depression Stigma Scale (DSS). This is a 9-item self report questionnaire to measure the personal stigma towards depression. It has 5-point Likert scale tanging from strongly disagree (1) and strongly agree (5). It had test-retest reliability of 0.71 and internal consistency of 0.76 (Griffiths KM et al. 2004)
help-seeking intentions | Through the study completion (pre and post-intervention), an average of one month
  The General Help-Seeking Questionnaire (GHSQ) has been developed to measure help-seeking intentions from different sources (friend, parent, mental health professional, and others) and is divided into personal-emotional problems and suicidal thoughts. The instrument consists of 10 items repeated twice for each part, measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). One question is stated as "I would not seek help from anyone" and is reverse scored. Higher scores on this scale indicate more help-seeking. The GHSQ has shown good psychometric properties: Cronbach's alpha = 0.70, and test-retest of 0.86 for personal-emotional problems, and Cronbach's alpha = 0.83, and test-retest of 0.88 for suicidal thoughts (Wilson CJ et al. 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Amsalem, MD, Study Director — Columbia University and NYSPI
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amsalem D, Martin A. Reducing depression-related stigma and increasing treatment seeking among adolescents: randomized controlled trial of a brief video intervention. J Child Psychol Psychiatry. 2022 Feb;63(2):210-217. doi: 10.1111/jcpp.13427. Epub 2021 Apr 6. PMID 33821507